CLINICAL TRIAL: NCT06018350
Title: Improving Medication Adherence in Chronic Rheumatic Diseases
Brief Title: Medication Adherence in Rheumatic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00108618
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Chronic Rheumatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Clinicians in this arm will be trained to conduct the adherence intervention in general rheumatology clinic with all follow up patients with a chronic rheumatic disease.
  Patients seen by these clinicians will contribute to the outcome data collection.
  Interventions: Behavioral: Clinician-led adherence intervention

INTERVENTIONS:
Behavioral: Clinician-led adherence intervention — The clinician will review real time pharmacy refill data during clinic and use effective communication techniques to discuss adherence with the patient

SUMMARY:
The investigators will pilot test a clinician-led intervention to improve medication adherence in general rheumatology clinic across a spectrum of rheumatic diseases. The study will assess feasibility, acceptability, and fidelity, and explore signal for improved medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* all providers at Southpoint Rheumatology All patients with a rheumatic disease diagnosis currently prescribed at least one rheumatic medication will be included in the analysis

Exclusion Criteria:

* new patients, those who are not prescribed any rheumatic disease medications, or do not have available pharmacy refill data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Sun, MD, MS, Principal Investigator — Duke Health
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinician-led Adherence Intervention - Clinicians: Clinicians in this arm will be trained to conduct the adherence intervention in general rheumatology clinic with all follow up patients with a chronic rheumatic disease.
  Patients seen by these clinicians will contribute to the outcome data collection.
  Clinician-led adherence intervention: The clinician will review real time pharmacy refill data during clinic and use effective communication techniques to discuss adherence with the patient
- Clinician-led Adherence Intervention - Patients: Patients seen by these clinicians will contribute to the outcome data collection.
  Clinician-led adherence intervention: The clinician will review real time pharmacy refill data during clinic and use effective communication techniques to discuss adherence with the patient
Period: Overall Study
Arm/Group | Clinician-led Adherence Intervention - Clinicians | Clinician-led Adherence Intervention - Patients
Started | 6 | 96
Completed | 6 | 96
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinician-led Adherence Intervention - Clinicians | Clinician-led Adherence Intervention - Patients | Total
Number analyzed (Participants) | 6 | 96 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data not collected on clinicians.
  years
    number analyzed (Participants) | 0 | 96 | 96
    (all) |  | 54 (17) | 54 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 81 | 83
  Male | 4 | 15 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 6 | 91 | 97
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 31 | 31
  White | 5 | 57 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 6 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 96 | 102

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility as Measured by Number of Providers Agreeing to Participate
Time Frame: 4 weeks
Population: Clinicians approached for study participation.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician-led Adherence Intervention - Clinicians
Number analyzed (Participants) | 6
Participants | 6

2. Primary Outcome: Intervention Feasibility as Measured by the Feasibility of Intervention Measure (FIM)
Description: Provider survey based on the Feasibility of Intervention Measure, scores range from 1-5, where 5 is most feasible.
Time Frame: 4 weeks
Population: Data not collected on patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician-led Adherence Intervention - Clinicians
Number analyzed (Participants) | 6
score on a scale | 4.60 (0.58)

3. Primary Outcome: Intervention Feasibility as Measured by Percent of Visits With EMR Documentation of Providers Reviewing Refills
Description: Calculated for the full population, not per participant.
Time Frame: 4 weeks
Measure: Number; unit: percentage of visits
Units Other Than Participants: Visits
Arm/Group | Clinician-led Adherence Intervention - Patients
Number analyzed (Participants) | 96
Number analyzed (Visits) | 96
percentage of visits | 65.0

4. Secondary Outcome: Intervention Acceptability as Measured by the Acceptability of Intervention Measure (AIM)
Description: Provider survey based on the Acceptability of Intervention Measure, scores range from 1-5, where 5 is most acceptable.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician-led Adherence Intervention - Clinicians
Number analyzed (Participants) | 6
score on a scale | 4.30 (0.64)

5. Secondary Outcome: Intervention Acceptability as Measured by the Percentage of Patients Who Report a Positive Feeling After Having an Adherence Conversation With Their Providers
Description: Patient survey will be administered following provider visit.
Time Frame: 4 weeks
Population: Patients who completed the survey.
Measure: Number; unit: percentage of patients
Arm/Group | Clinician-led Adherence Intervention - Patients
Number analyzed (Participants) | 42
percentage of patients | 90.0

6. Secondary Outcome: Fidelity as Measured by the Number of Participants With Clinicians Conducting the Intervention Components of Reviewing Pharmacy Refills and Using Effective Communication Strategies
Description: This was collected using a EMR Smartphrase where clinicians documented whether they reviewed pharmacy refill data or discussed adherence with patients.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician-led Adherence Intervention - Patients
Number analyzed (Participants) | 96
Participants | 62

7. Secondary Outcome: Fidelity as Measured by the Number of Participants With EMR Documentation of Completing the Intervention Components of Reviewing Pharmacy Refills and Using Effective Communication Strategies
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician-led Adherence Intervention - Patients
Number analyzed (Participants) | 96
Participants | 62

8. Secondary Outcome: Change in MPR (Medication Possession Ratio) as a Percentage for the Entire Sample
Description: MPR is calculated by dividing the number of days all patients were covered by medication by the total number of days in the observation period. This is multiplied by 100 to present a percent change for the entire sample.
Time Frame: Baseline to 3 months
Measure: Number; unit: percentage of change
Arm/Group | Clinician-led Adherence Intervention - Patients
Number analyzed (Participants) | 96
percentage of change | 11.0
Statistical Analysis 1: Comparison: Clinician-led Adherence Intervention - Patients; Test type: Other; p = 0.002, McNemar

9. Other Pre Specified Outcome: Change in MPR (Medication Possession Ratio) as a Percentage
Description: MPR is calculated by dividing the number of days a patient is covered by medication by the total number of days in the observation period. This is multiplied by 100 to present a percent change.
Time Frame: Baseline to 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Clinician-led Adherence Intervention - Clinicians | Clinician-led Adherence Intervention - Patients
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/96
Other Adverse Events (participants affected / at risk) | 0/6 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT06018350/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT06018350/ICF_000.pdf